CLINICAL TRIAL: NCT05449093
Title: Gingival Crevicular Fluid Galectin-3 and Interleukin-1beta Levels in Stage 3 Periodontitis With Grade B and C.
Brief Title: GCF Galectin-3 and Interleukin-1beta Levels in Periodontitis.
Status: Completed | Type: Observational
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Beral Afacan, Associate Professor, Aydin Adnan Menderes University
Other Study IDs: bafacan0922
Record Dates: First submitted 2022-07-04; First posted 2022-07-08 (Actual); Last update posted 2022-07-08 (Actual); Status verified 2022-07

CONDITIONS: Periodontitis; Periodontal Inflammation
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Gingival crevicular fluid
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Stage 3 Grade C Periodontitis: Generalized stage 3 periodontitis patients had interproximal clinical attachment loss ≥ 5 mm at 30 % of the teeth or more. Care was taken to ensure that clinical attachment loss was caused by periodontal causes. These patients had also radiographic bone loss extending to the mid-third of the root or beyond and probing depth ≥ 6 mm at 30 % of the teeth or more as well as Class II-III furcation involvement. The grade of periodontitis was estimated with indirect evidence of progression through % of bone loss/age. Radiographic bone loss of each natural tooth was assessed by using the panoramic radiograph. The tooth showing the most extensive bone loss was determined and % of bone loss/age were calculated. If this value was higher than 1.0, the patients were assigned to grade C.
  Interventions: Other: Periodontal clinical measurements and gingival crevicular fluid sampling
- Stage 3 Grade B Periodontitis: Generalized stage 3 periodontitis patients had interproximal clinical attachment loss ≥ 5 mm at 30 % of the teeth or more. Care was taken to ensure that CAL was caused by periodontal causes.These patients had also radiographic bone loss extending to the mid-third of the root or beyond and probing depth ≥ 6 mm at 30 % of the teeth or more as well as Class II-III furcation involvement. The grade of periodontitis was estimated with indirect evidence of progression through % of bone loss/age. Radiographic bone loss of each natural tooth was assessed by using the panoramic radiograph. The tooth showing the most extensive bone loss was determined and % of bone loss/age were calculated. When this value was between 0.25 and 1.0, patients were included in grade B.
  Interventions: Other: Periodontal clinical measurements and gingival crevicular fluid sampling
- Gingivitis: Gingivitis patients showed probing depth ≤ 3 mm with bleeding on probing ≥ 30 % in the entire mouth as well as no interproximal clinical attachment loss or radiographic bone loss.
  Interventions: Other: Periodontal clinical measurements and gingival crevicular fluid sampling
- Periodontal Health: Periodontally healthy individuals in the control group had an intact periodontium or a reduced periodontium (without detectable interproximal clinical attachment loss or radiographic bone loss) in a non-periodontitis patient. In this group, probing depth was ≤ 3 mm and bleeding on probing was < 10 % in the whole mouth.
  Interventions: Other: Periodontal clinical measurements and gingival crevicular fluid sampling

INTERVENTIONS:
Other: Periodontal clinical measurements and gingival crevicular fluid sampling — Periodontal clinical meaurements including the probing depth, clinical attachment loss, the dichotomous recording (present/absent) of bleeding on probing, gingival index, and the plaque index at six sites (distobuccal, buccal, mesiobuccal, distopalatinal/lingual, palatinal/lingual, mesiopalatinal/lingual) on all teeth, except third molars, were performed using manuel periodontal probe.
  Standardized absorbent paper strips were used for gingival crevicular fluid sampling. A sterile paper strip was gently inserted into the gingival sulcus/periodontal pocket until mild resistance was felt and were kept in place for 30 seconds. The absorbed fluid volume was measured by a precalibrated electronic device.

SUMMARY:
This study aims to evaluate gingival crevicular fluid Galectin-3 and Interleukin-1beta levels in different grades (B and C) of stage 3 periodontitis, concurrently, and also to investigate their discriminative efficiencies in periodontal diseases. A total of 80 systemically healthy and non-smoker individuals, 20 stage 3 grade C periodontitis 20 stage 3 grade B periodontitis, 20 gingivitis and 20 periodontally healthy were enrolled. Clinical periodontal parameters were recorded and GCF Galectin-3 and interleukin-1 beta total amounts were measured by ELISA. Receiver operating characteristics curve was used for estimating the area under the curve.

DETAILED DESCRIPTION:
A total of 80 systemically healthy and non-smoker individuals, 20 stage 3 grade C periodontitis 20 stage 3 grade B periodontitis, 20 gingivitis and 20 periodontally healthy were enrolled.

Periodontal clinical measurements including the probing depth, clinical attachment loss, the dichotomous recording (present/absent) of bleeding on probing, gingival index, and the plaque index at six sites (distobuccal, buccal, mesiobuccal, distopalatinal/lingual, palatinal/lingual, mesiopalatinal/lingual) on all teeth, except third molars, were performed by a graded periodontal probe.

According to the diagnostic criteria proposed by the 2017 International Workshop on the Classification of Periodontal and Peri-implant Diseases and Conditions18 participants were classified into four distinct groups based on their periodontal conditions: 1) 20 patients with generalized stage 3 grade C periodontitis; 2) 20 patients with generalized stage 3 grade B periodontitis; 3) 20 patients with gingivitis; and 4) 20 periodontally healthy individuals.

Gingival crevicular fluid was sampled from the buccal aspects of two non-adjacent interproximal sites in single-rooted teeth. Standardized absorbent paper strips were used for sampling. In periodontitis groups, samples were taken from two deepest pockets of single-rooted teeth. Samples were obtained from the sites with visible signs of inflammation in patients with gingivitis and without bleeding on probing in the healthy controls. The absorbed fluid volume was measured by a precalibrated electronic device.

Galectin-3 and interleukin-1 beta levels in gingival crevicular fluids samples were measured by the ELISA via commercial kits in line with the manufacturer's guidelines. Protein concentrations were calculated from the standard curve. Gingival crevicular fluid results for two analytes were expressed as total amounts at two samples per sampling time.

Normality of the data was checked by Shapiro Wilk's normality test. Comparisons of clinical parameters and gingival crevicular fluids biomaker levels among the study groups were performed using Kruskal-Wallis test and Dunn's test (with Bonferroni correction) was used to pairwise comparisons for non-normally distributed variables. Receiver operating characteristic (ROC) curves were constructed to assess the ability of two analytes for diagnosis of periodontitis. Statistical significance was considered at p< 0.05 for all the tests.

ELIGIBILITY:
Inclusion Criteria:

* Non-smokers with no history of smoking (determined by self-reporting)
* Individuals who had at least 20 teeth (excluding third molars)

Exclusion Criteria:

* Patients with diagnosed medical illness such as diabetes mellitus, rheumatoid arthritis, cardiovascular diseases, immunological diseases.
* Patients who under any medication including immunosuppressants, steroids, non-steroidal anti-inflammatory drugs, antibiotics, antiepileptic drugs, calcium channel blockers, beta-blockers, anticoagulants, hormonal contraceptives and nutritional supplements within the past 6 months, topical antiseptic solutions in the last 3 months.
* Pregnant and lactating women
* Individuals who had orthodontic appliances or removable partial dentures
* Individuals who had undergone professional teeth cleaning within the past year

Ages: 25 Years to 52 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: A total of 80 systemically healthy and non-smoker individuals (36 males and 44 females) aged 25-52 years were consecutively included.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2019-02-21 (Actual); Primary Completion 2019-08-23 (Actual); Study Completion 2019-09-02 (Actual)

PRIMARY OUTCOMES:
Gingival crevicular fluid Galectin-3 levels | 24 hours after clinical periodontal measurements
  ng
Gingival crevicular fluid interleukin-1 beta levels | 24 hours after clinical periodontal measurements
  pg

CONTACTS AND LOCATIONS:
Overall Officials: Beral Afacan, Principal Investigator — Aydin Adnan Menderes University; Gülnur Emingil, Study Director — İzmir Ege University; Harika Atmaca İlhan, Principal Investigator — Manisa Celal Bayar University; Timur Köse, Principal Investigator — İzmir Ege University
Locations (1):
- Adnan Menderes University, Faculty of Dentistry, Department of Periodontology, Aydin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No